CLINICAL TRIAL: NCT07249216
Title: Identification of Molecular Signals in Vitreous Humor Associated With Suboptimal Response to VEGF Inhibition in nAMD Within a Clinical Trial Setting
Brief Title: Identification of Molecular Signals in Vitreous Humor Associated With Suboptimal Response to Vascular Endothelial Growth Factor (VEGF) Inhibition in Neovascular Age-related Macular Degeneration (nAMD) Within a Clinical Trial Setting
Acronym: M-VIVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Gemmy Cheung Chui Ming, Professor, Singapore Eye Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2025-0319
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — faricimab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ranibizumab (Other)
  Interventions: Drug: Ranibizumab
- Faricimab (Other)
  Interventions: Drug: Faricimab; Drug: Ranibizumab

INTERVENTIONS:
Drug: Faricimab — All study eyes will start on the intravitreal ranibizumab loading phase, with the initial injection given within two weeks of the screening visit and overall of x 3 monthly injections.
  At week 12, patients will be evaluated for their response following the loading phase. Patients who show an absence of IRF, absence of or ≤100µm subretinal fluid (SRF), and no new hemorrhage will be categorized as good responders and will continue with four further monthly intravitreal ranibizumab. Suboptimal responders (defined as the presence of subretinal fluid > 100 µm, any intraretinal fluid (IRF), or a new hemorrhage) will switch to four doses of monthly intravitreal faricimab.
  Arms: Faricimab
Drug: Ranibizumab — All study eyes will start on the intravitreal ranibizumab loading phase, with the initial injection given within two weeks of the screening visit and overall of x 3 monthly injections.
  At week 12, patients will be evaluated for their response following the loading phase. Patients who show an absence of IRF, absence of or ≤100µm SRF, and no new hemorrhage will be categorized as good responders and will continue with four further monthly intravitreal ranibizumab. Suboptimal responders (defined as the presence of subretinal fluid > 100 µm, any intraretinal fluid (IRF), or a new hemorrhage) will switch to four doses of monthly intravitreal faricimab.

SUMMARY:
Neovascular age-related macular degeneration (nAMD), also called wet AMD, can cause serious vision loss. While anti-VEGF (anti Vascular Endothelial Growth Factor) treatments such as ranibizumab help many patients, about 20 40% have a suboptimal response. In this study, the investigators want to identify other factors (beyond VEGF) that might be driving the disease in these non-responding patients. By looking at samples from inside the eye (vitreous humor) and comparing "good responders" to "suboptimal responders", the investigators hope to find potential new treatment approaches or biomarkers for nAMD.

DETAILED DESCRIPTION:
Neovascular age-related macular degeneration (nAMD) is a leading cause of severe vision loss worldwide. Although intravitreal anti-VEGF injections have markedly improved outcomes, 20-40% of patients show a suboptimal response, indicating the involvement of additional molecular pathways. This study investigates whether profiling the vitreous humor can reveal alternative angiogenic pathways-beyond VEGF-that drive persistent disease. If such pathways are identified, switching from anti-VEGF monotherapy (ranibizumab) to a bispecific anti-VEGF/anti-Ang2 agent (faricimab) may improve disease control and provide better vision outcomes for patients with inadequate response to standard therapy.

Additionally, the dosage regimens (monthly injections over 24 weeks), and selection of treatment-naïve nAMD patients will minimize confounding variables. This approach ensures a clear comparison between good responders and suboptimal responders. By correlating clinical/imaging outcomes with vitreous biomarker profiles, the investigators aim to develop personalized treatment strategies for nAMD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 50 years old at the time of informed consent
2. Willing and able to provide informed consent
3. Willingness and ability to comply with all scheduled visits and study procedures
4. Female subjects must be of non-childbearing potential or show a negative pregnancy test at screening and must agree to use appropriate methods of contraception during the study and for one month after the last dose.
5. Confirmed diagnosis of symptomatic nAMD based on optical coherence tomography (OCT), fluorescein fundus angiography (FFA), and indocyanine green angiography (ICG-A)
6. nAMD characteristics:

   1. Subfoveal CNV/PCV
   2. Juxtafoveal/extrafoveal CNV/PCV with a subfoveal component related to the exudative activity.
7. Treatment naïve- NO previous treatment with intravitreal anti-VEGF agents, regardless of the indication, NO previous thermal laser in the macular region, or verteporfin photodynamic therapy (vPDT), regardless of indication
8. BCVA of 24-78 letters as measured by an Early Treatment Diabetic Retinopathy Study (ETDRS) chart (Snellen equivalent 20/32-20/320)

Exclusion Criteria:

1. CNV or retinal exudation due to causes other than typical AMD, such as vitelliform dystrophy, ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, or uveitis
2. Active intraocular inflammation or suspected or active intraocular or periocular infection (eg, infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis) in either eye at Baseline
3. Any history or evidence of a concurrent intraocular condition in the study eye, including retinal diseases other than neovascular AMD, that, in the judgment of the Investigator, could either require medical or surgical intervention during the course of the study to prevent or treat visual loss that might result from that condition or that limits the potential to gain visual acuity upon treatment with the investigational product

   * History of cataract surgery within 6 months prior to recruitment
   * Cataract surgery during the study period is not permitted.
4. Retinal pigment epithelium (RPE) rip/tear in the study eye at Baseline
5. Current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to Baseline
6. History of rhegmatogenous retinal detachment, stage 3/4 macular hole, or any retinal break unless adequate repair has been performed
7. History of the following in the study eye:

   * Previous pars plana vitrectomy
   * Previous photodynamic therapy (PDT)
   * Intraocular or refractive surgery within the 6 months period prior to Baseline
   * Previous penetrating keratoplasty or vitrectomy
   * Previous pan retinal photocoagulation
   * Previous submacular surgery or macular laser treatment
8. Uncontrolled glaucoma or ocular hypertension in the study eye defined as intraocular pressure (IOP) > 25 mmHg on medication or according to the investigator's judgment at baseline
9. Intra- or periocular use of corticosteroids in the study eye during the 6-month period prior to baseline:

   1. Use of topical ocular corticosteroids in the study eye for 60 or more consecutive days within the 90-day period prior to baseline
   2. Use of systemic corticosteroids for 30 or more consecutive days within the 90 days prior to baseline, with the exception of low stable doses of corticosteroids (defined as ≤10 mg prednisolone or equivalent dose used for 90 days or more). Inhaled, nasal or dermal steroids are also permitted
10. Previous therapeutic radiation near the region of the study eye
11. History of a medical condition (disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding) that, in the judgment of the investigator, would preclude scheduled study visits, completion of the study, or a safe administration of the investigational product
12. History of hypersensitivity to any component of the test article or clinically relevant sensitivity to fluorescein dye (or indocyanine green), as assessed by the Investigator
13. Participation in an investigational drug, biologic, or device study within 30 days or the duration of 5 half-lives of the investigational product (whichever is longer) prior to baseline Note: observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary
14. Systemic anti-vascular endothelial growth factor (VEGF) therapy within the 90-day period prior to baseline
15. Stroke or myocardial infarction in the 90-day period prior to baseline
16. Uncontrolled blood pressure defined as a systolic value ≥ 180 mmHg and/or diastolic value ≥ 100 mmHg at screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Difference in vitreous biomarker concentrations between responders and non-responders | 24 weeks
  Comparison of inflammatory and angiogenic biomarkers in vitreous humor measured at baseline, week 12, and week 24

SECONDARY OUTCOMES:
Change in concentration of inflammatory and angiogenic biomarkers in vitreous humor from baseline to week 24 (including IL-6, IL-8, MCP-1, TNF-α, VEGF-A, PlGF, ANG-2, MMP-2, MMP-9, and complement pathway proteins) | 24 weeks
  Picograms per milliliter (pg/mL)
Proportion of eyes classified as suboptimal responders at Week 12 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre/Singapore Eye Research Institute, Singapore, Singapore